CLINICAL TRIAL: NCT06182267
Title: A Randomized, Crossover, Controlled, Maximal Use Study to Determine the Pharmacokinetics of L-arginine After Exaggerated Oral Use of COL101 in Healthy Adult Subjects
Brief Title: Maximal Use Study to Determine the Pharmacokinetics of L-arginine After Exaggerated Oral Use of COL101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2023-10-TKL-GPS-JM
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Caries,Dental
Keywords: arginine
MeSH Terms: conditions — Dental Caries | interventions — Arginine; Sodium Fluoride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Experimental): toothpaste containing 8% L-arginine
  Interventions: Drug: L Arginine; Drug: Sodium Fluoride
- Group II (Active Comparator): toothpaste containing 0.24% sodium fluoride
  Interventions: Drug: L Arginine; Drug: Sodium Fluoride

INTERVENTIONS:
Drug: L Arginine — toothpaste
Drug: Sodium Fluoride — toothpaste

SUMMARY:
Pharmacokinetic (PK) study of L-arginine after exaggerated oral use of the novel dentifrice product COL101 after repeated daily applications in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 - 65 years of age;
* In good health as determined by medical history, physical and dental examination, vital signs and clinical laboratory safety assessment;
* Agree to delay any elective dentistry including dental prophylaxis until the study has been completed;
* Agree to refrain from supplements containing arginine throughout the duration of the study;
* In the case of females of childbearing potential (unless surgically sterilized [hysterectomy, bilateral oophorectomy, tubal ligation] or are postmenopausal for at least 12 months), are using one acceptable form of birth control (oral/implant/injectable/transdermal contraceptives, intrauterine device (IUD), condom with spermicide, diaphragm with spermicide, partner's vasectomy). Abstinence or vasectomies are acceptable if the female subject agrees to implement an acceptable form of birth control if her lifestyle/partner changes;
* For females of childbearing potential, have a negative serum pregnancy test (SPT) at the Screening visit and a negative urine pregnancy test (UPT) on Day -2 prior to randomization, and agree to submit to a SPT at the end of study (EOS) visit;
* Are free of any systemic or dermatologic disorder, which, in the opinion of the Principal Investigator (PI), will interfere with the study results or increase the risk of adverse events (AEs); and
* Read, understand, and provide signed informed consent.

Exclusion Criteria:

* A female who is pregnant, plans to become pregnant during the study, or is breastfeeding a child;
* Are actively being treated for periodontitis, gingivitis or caries;
* Have severe periodontal disease, as characterized by purulent exudates, generalized mobility, or severe recession;
* Any clinically significant central nervous system, cardiac, pulmonary, renal, gastrointestinal (GI), endocrinological, respiratory, or metabolic conditions (or history), or other pathological or physiological conditions, that might interfere with the study results in the investigator's opinion;
* Any condition which, in the investigator's opinion, puts the subject at significant risk, could confound the study results, or may interfere significantly with the subject's participation in the study;
* Have known or suspected allergies to oral care products, toothpaste, or ingredients in toothpaste;
* Immunization within 10 days of Day 1;
* Anticipated need for surgery or hospitalization during the study;
* Consumed alcohol within 48 hours prior to Day 1 or refuses to abstain from alcohol throughout the duration of the study;
* History of heavy smoking (i.e., more than 10 cigarettes a day or the tobacco/nicotine equivalent) within 3 months of screening or refuses to abstain from tobacco or nicotine-containing products throughout the duration of the study;
* Consumed caffeine (i.e., coffee, tea, caffeinated soda, chocolate) within 48 hours prior to Day 1 or refuses to abstain from caffeine throughout the duration of the study;
* Donation or loss of blood (excluding volume drawn at screening) of ≥ 450 mL within 3 months of Day 1;
* Active or lifetime infection (e.g., negative test for human immunodeficiency virus (HIV) and hepatitis, and no history of tuberculosis and syphilis) or a history of severe infection during the 30 days prior to screening;
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment;
* Is unwilling or unable to refrain from using prescription medications for 30 days prior to Day 1 or over the counter medications, herbal preparations, and supplements for 14 days prior to Day 1 (excluding permitted forms of contraception and occasional use of acetaminophen [up to 2 g in 24 hours]);
* Inability or unlikeliness of the subject to comply with the dose schedule and study evaluations, in the opinion of the investigator;
* Is currently participating in any clinical trial;
* Has received any investigational drug(s) within 30 days or 5 half-lives, whichever is longer, prior to study Day 1;
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data;
* Inability of the subject (or legally authorized representative) to comprehend the electronic informed consent form (eICF) or unwillingness to sign the eICF; and/or
* Subject meets eligibility criteria, but study is filled

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Arginine in blood | Day 1 for 24 hours
  Measurement of arginine in blood after oral brushing
Arginine in blood | Day 7 for 24 hours
  Measurement of arginine in blood after oral brushing
Arginine in blood | Day 10 for 24 hours
  Measurement of arginine in blood after oral brushing
Arginine in blood | Day 16 for 24 hours
  Measurement of arginine in blood after oral brushing

CONTACTS AND LOCATIONS:
Overall Officials: Irina Krause, RN, MSN, Study Director — TKL
Locations (1):
- TKL Research, Inc, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No